CLINICAL TRIAL: NCT06798844
Title: Spinal Cord Stimulation for Freezing of Gait in Parkinson's Disease
Acronym: SCSforFOG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S69667; CIV-24-10-049614 (Registry Identifier: Eudamed); 402173 (Registry Identifier: Single Identification Number (SIN))
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Freezing of Gait; Parkinson Disease
Keywords: Spinal Cord Stimulation; Freezing of Gait; Parkinson disease
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Sham-controlled randomized double-blinded cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the patient and assessors will be blinded to the SCS paradigm during the core trial. Upon the patient's completion of the core trial (the 3-week trial stimulation period) and after blinded assessment of all videos, the investigator will be unblinded to the patient's treatment response to evaluate the effect of SCS on FOG. This information is critical for determining, in consultation with the patient, whether to proceed with the implantation of a definitive internal neurostimulator or to remove the trial electrode. It is important to note that, as previously stated, the investigator and assessors remain blinded to the patient's assigned SCS paradigm throughout the whole core trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PD patients with refractory FOG (Experimental): 29 PD patients with refractory FOG will receive a 3-week SCS trial with an implanted lead connected to an external stimulator, during which two SCS paradigms (one with and one without paraesthesia) and a sham paradigm will be compared. If a clinically relevant improvement in FOG or gait is perceived during the external trial stimulation, the participant will receive a permanent implanted neurostimulator.
  Interventions: Device: Spinal Cord Stimulation
- Control group 1: SCS patients without PD (Other): ± 15 patients without PD who received SCS for FBSS outside research settings.
  To evaluate the secondary exploratory outcome on spinal cord electrophysiology in PD freezers, two control groups of SCS patients treated for approved indications outside research settings will be included. This allows for an exploratory, non-blinded, and non-randomized comparison of spinal cord electrophysiological characteristics between patients with PD and FOG (intervention group), without PD (control group 1) and with PD without FOG (control group 2).
  Interventions: Other: Spinal electrophysiological recordings
- Control group 2: SCS patients with PD, without FOG (Other): Max. 5 patients with PD without FOG who received SCS for FBSS outside research settings.
  To evaluate the secondary exploratory outcome on spinal cord electrophysiology in PD freezers, two control groups of SCS patients treated for approved indications outside research settings will be included. This allows for an exploratory, non-blinded, and non-randomized comparison of spinal cord electrophysiological characteristics between patients with PD and FOG (intervention group), without PD (control group 1) and with PD without FOG (control group 2).
  Interventions: Other: Spinal electrophysiological recordings

INTERVENTIONS:
Device: Spinal Cord Stimulation — SCS is an established treatment for chronic neuropathic pain and the implantation procedure in this study follows the conventional clinical approach. Under local anaesthesia, a lead electrode is positioned in the spinal epidural space at the Th8-Th10 vertebral levels. The electrode is then connected to an external stimulator (implantable pulse generator, IPG), used for the 3-week external trial stimulation. Upon completion of the core trial, the electrode may either be removed or connected to an internal IPG, after extensive counselling and dependent on the FOG outcome and patient's preference. A subsequent long-term open label phase will evaluate the long-term efficacy and safety of SCS on FOG, with a follow-up period of six months. Electrophysiological recordings of the dorsal spinal cord will be conducted at the end of the external trial stimulation and at the 6-month follow-up.
  Other Names: Medtronic Inceptiv neurostimulator
  Arms: PD patients with refractory FOG
Other: Spinal electrophysiological recordings — The sole purpose of the control groups in this study, is to facilitate the interpretation of spinal cord electrophysiological characteristics in PD freezers by providing a comparison with individuals without the condition.
  Arms: Control group 1: SCS patients without PD; Control group 2: SCS patients with PD, without FOG

SUMMARY:
Freezing of gait (FOG) is a severely disabling gait disorder in Parkinson's disease (PD). Its poor response to current therapies reflects the shortfall in current knowledge on its exact pathophysiology. Case series suggest a therapeutic promise of spinal cord stimulation (SCS) for FOG, but double-blind randomised controlled trials with reliable FOG assessments are lacking.

This randomised, double-blind, placebo-controlled cross-over trial aims to define the outcome, safety, optimal stimulation paradigm and underlying mechanism of SCS for FOG in PD, by exploring both clinical and neurophysiological parameters.

Twenty-nine PD patients with refractory FOG will receive an implanted SCS lead connected to an external trial stimulator. During a 3-week trial, 3 stimulation paradigms will be tested in random order, including one sham paradigm. SCS outcome on FOG will be evaluated through wearable accelerometers, self-reported questionnaires and a FOG-provoking protocol at home. Spinal electrophysiological recordings will compare neural properties between PD patients with and without FOG and evaluate intra-patient differences (e.g., on/off medication, DBS states). In patients with deep brain stimulation (DBS) including BrainSense technology, the effect of SCS on pathological beta oscillations in the STN will be explored. A subsequent long-term open-label phase will be conducted in those patients who desire a definitive implanted stimulator.

This project will provide new insights into the pathophysiology of FOG, pave the way for SCS implementation in clinical practice and enhance future patient selection.

DETAILED DESCRIPTION:
Freezing of gait (FOG) is a severely disabling gait disorder in Parkinson's disease (PD). FOG leads to falls, anxiety and loss of independence and heavily affects quality of life (QoL). The incidence of FOG increases from 38% in the first 5 years following diagnosis to 65-80% in advanced stages. FOG is a therapeutic challenge, as it often responds poorly to (dopaminergic) pharmacotherapy or deep brain stimulation (DBS) of the subthalamic nucleus (STN) or internal pallidum. Likewise, rehabilitation strategies such as gait training achieve small and short term effects at best. The therapeutic response of FOG is far more complex and variable than that of other PD motor symptoms. This reflects the current shortfall in knowledge about FOG pathophysiology, which has drastically impeded adequate therapy development. Furthermore, objective and reliable FOG assessments are challenging and therefore still rarely implemented in clinical trials, limiting the interpretation of the findings. However, recent insight into the underlying mechanisms has resulted in a growing body of literature suggesting a therapeutic promise of spinal cord stimulation (SCS) for FOG.

Spinal cord stimulation is an invasive technique in which specific neuronal circuits are stimulated electrically through spinal epidural electrodes. The stimulation settings can be adjusted to achieve a therapeutic effect, often by eliciting paraesthesia. SCS has been applied mostly in patients with refractory neuropathic pain. Serendipitously, PD patients who underwent SCS to treat comorbid neuropathic pain also noticed a beneficial effect on FOG. This finding led to SCS being further investigated as a therapy for FOG, but despite the encouraging results in animal studies, studies in humans are limited to case reports and series with inconsistent results. Randomised, double-blinded, high-quality trials in large cohorts are much needed for translation to clinical use. Correct blinding in SCS studies was historically impeded by stimulation-induced paraesthesia. However, recent innovations in SCS devices now enable paraesthesia-free stimulation and spinal cord electrophysiology recordings, creating new opportunities for research and trial design.

In addition to the small sample sizes and lack of randomisation and blinding, currently published reports on SCS for FOG lack clear clinical phenotyping of freezing and many also fail to use objective, reliable FOG assessments. Moreover, much remains unknown about the effect of SCS on spinal cord and STN electrophysiology and about optimal stimulation paradigms.

This sham-controlled randomized double-blinded cross-over study aims to define the outcome, safety, optimal stimulation paradigm and underlying mechanism of SCS for FOG in PD patients. Twenty-nine patients will receive a 3-week SCS trial with an implanted lead connected to an external stimulator, during which two SCS paradigms (one with and one without paraesthesia) and a sham paradigm will be compared:

1. Tonic SCS (paraesthesia-eliciting)
2. DTM SCS (paraesthesia-free)
3. Sham SCS (stimulation off)

The three SCS paradigms will be evaluated for 5 days each in a randomised order, split by a 2-day wash-out. SCS outcome on FOG will be evaluated through a wearable accelerometer, questionnaires and a FOG-provoking protocol at home. During this FOG-provoking protocol, participants have to perform 4 different tasks:

1. Timed Up and Go test;
2. One minute of 360° turns in place, alternating the direction after each turn;
3. Bathroom task, where patients have to walk 2m, enter the toilet through the doorway, turn around there and return to the starting position;
4. Clearing the table, where patients need to set and clear the table with 2 plastic plates and cups. Starting and ending point is at 2m away from the table. During the task, they are also required to move the chairs in place.

The first two tasks will be executed twice, once while dual-tasking (serial-3 subtractions) and once without. Patients are allowed to use a walking aid if necessary to complete the protocol. Each FOG-protocol is conducted both in off-meds (≥ 12h withdrawal) and on-meds (±1h after intake) conditions. The entire protocol is videorecorded and annotated afterwards to determine percentage time frozen (%TF) and characterisation of FOG. During the FOG-protocol, the participant will wear 5 intertial measurement units to quantify gait parameters. In patients with DBS including BrainSense technology, we will explore the effect of SCS on pathological beta oscillations in the STN.

Upon completion of the core trial, participants who exhibit a clinically relevant improvement in freezing or gait will receive a permanent implanted neurostimulator and continue into the long-term open-label phase. In participants who do not perceive a clinically relevant FOG improvement from SCS during the core trial, the trial electrode is removed. Six months following either implantation of the permanent neurostimulator or removal of the trial electrode, long-term therapeutic efficacy and safety of SCS for FOG will be assessed and compared between patients who received permanent SCS and those who did not. In addition, electrophysiological recordings of the dorsal spinal cord will be conducted at the end of the external trial stimulation and at the 6-month follow-up. These electrophysiological signal characteristics will be compared to two control groups of patients who received an Inceptiv SCS system outside research settings for approved indications (one group without PD, one group with PD but without FOG).

To conclude, this study will provide new insights into the pathophysiology of FOG, pave the way for SCS implementation in clinical practice and enhance future patient selection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD in accordance with the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease
* Optimal medical or DBS management for FOG, as evaluated by a movement disorder neurologist and programming expert. Stable PD medication and/or DBS settings for ≥ 1 month prior to baseline assessment and no changes are expected for the next 8 weeks
* Self-reported FOG severity of ≥ 1 FOG episode per day, based on NFOG-Q items 1 and 2
* Presence of FOG during in-hospital clinical assessment consisting of 3 FOG-provoking tasks, in the on-medication state
* Able to walk 10 meters unassisted without a walking aid (use of a cane is allowed)
* Able to understand study requirements and provide consent
* Age 40-79 years inclusive

Exclusion Criteria:

* Presence of other severe neurological, psychiatric or other disorder that may impede assessment of outcomes
* Contra-indications to SCS surgery (e.g. epidural fibrosis, inability to safely discontinue anticoagulant drugs, allergy to implants, medically inoperable)
* Cognitive impairment (Montreal Cognitive Assessment (MOCA) <19/30)
* Chronic (>6m) severe (numeric rating scale >5/10) back or leg pain, or FBSS, as the antalgic effect of SCS could cloud our interpretations for its effect on FOG
* Duodopa pump or apomorphine injections
* Fall frequency >1x/day (this criterion comprises only 'actual falls', no 'near falls')
* Absence of FOG during preoperative at-home FOG-protocol, in on- or off-medication assessment
* Pregnancy, lactating or active pregnancy plans

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
FOG-provoking protocol | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  The total percentage time frozen (%TF) of all FOG manifestations across all gait tasks of the FOG-protocol performed in the off medication state, compared between the different SCS paradigms.

SECONDARY OUTCOMES:
Safety | 6 months
  Adverse event (AE) frequency, severity and causality
FOG-provoking protocol | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  The total %TF of all FOG manifestations across all gait tasks of the FOG-protocol performed in the on medication state, compared between the different SCS paradigms.
FOG-provoking protocol | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  The %TF in both off- and on medication states for the different FOG manifestations, and for each of the different gait tasks of the FOG-protocol, compared between the different SCS paradigms.
Changes in home-based gait function | Core-trial: 3 weeks
  Objective assessment of changes in gait quantity and quality during daily life at home, using biometric data collected by a wearable accelerometer throughout the core trial. Data will be compared across the different SCS paradigms to evaluate their impact on everyday gait performance.
Patient Global Impression of Improvement (PGI-I) | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  Single-item questionnaire to assess the patient's perception of improvement in symptom severity. The scale ranges from 1 to 7, where 1 indicates "very much improved," and 7 indicates "very much worse." It will be compared between the 3 SCS paradigms.
Changes in daily patient-reported FOG severity, falls and near-falls | Core-trial: 3 weeks
  During the core trial, participants have to answer 3 questions every evening using a patient diary:
  "How do you rate your freezing severity today (scale 0-10)?"; "How many times did you fall today?", "How many times did you nearly fall today?".
  These measures will be compared between the 3 SCS paradigms.
Change in Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III and part IV.6 | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  MDS-UPDRS part III: 19-item clinical examination to assess motor symptoms of PD; MDS-UPDRS part IV item 6: to assess painful dystonia in the off medication state.
  Scores will be compared between the 3 SCS paradigms.
Change in Numeric (Pain) Rating Scale (NRS) | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  Pain scales will be collected to correct for FOG improvement through a possible antalgic effect of SCS.
Change in Medication Quantification Scale (MQS) | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  Pain medication scales will be collected to correct for FOG improvement through a possible antalgic effect of SCS.
Patient satisfaction | Core-trial: 3 weeks
  At the end of the core trial, patients will be asked which paradigm they preferred and whether they desire stimulator implantation.
Change in New Freezing of Gait Questionnaire (NFOG-Q) | 6 months
  9-item questionnaire to assess the presence, frequency, and impact of FOG. Scores will be compared at the 6-month follow-up to baseline.
Change in Characterizing Freezing of Gait questionnaire (C-FOG) | 6 months
  35-item questionnaire to characterize situations and strategies that trigger or relieve FOG. Scores will be compared at the 6-month follow-up to baseline.
Change in Parkinson's Disease 39-Item Quality of Life Questionnaire (PDQ-39) | 6 months
  39-item questionnaire to assess quality of life in PD. Scores will be compared at the 6-month follow-up to baseline.
Change in Levodopa Equivalent Daily Dose (LEDD) | 6 months
  Standardized measure used to calculate the total daily dose of various PD medications in terms of their equivalent potency to levodopa. LEDD will be compared at the 6-month follow-up to baseline.
Change in Parkinson Anxiety Scale (PAS) | 6 months
  12-item questionnaire to assess anxiety symptoms in PD. Scores will be compared at the 6-month follow-up to baseline.
Change in Beck Depression Inventory (BDI) | 6 months
  21-item questionnaire to assess depressive symptoms. Scores will be compared at the 6-month follow-up to baseline.
Change in Rem Sleep Behaviour Disorder Screening Questionnaire (RBDSQ) | 6 months
  13-item questionnaire to assess symptoms of REM sleep behaviour disorder. Scores will be compared at the 6-month follow-up to baseline.
Change in SCales for Outcomes in PArkinson's disease - Autonomic Dysfunction (SCOPA-AUT) | 6 months
  23-item questionnaire to assess autonomic symptoms in PD. Scores will be compared at the 6-month follow-up to baseline.
Patient satisfaction | 6 months
  Two questions at 6 months after internal stimulator implantation (only in patients who receive internal stimulator):
  "Knowing what you know now, would you agree to have the same neurosurgical intervention again?"; "Would you recommend this neurosurgical intervention to another patient suffering from the same condition?"

OTHER OUTCOMES:
STN-LFP recordings | Core trial: day 7, 14 and 21 post-surgery. Long-term: at 6 months follow-up.
  (1) Changes in LFP spectrum (e.g. β activity) and (2) possible correlations with FOG alleviation, measured in patients with STN-DBS (Medtronic Percept PC) during the FOG-provoking protocol.
Spinal electrophysiological recordings | at 3 weeks and at 6 months
  Changes in spinal cord electrophysiological characteristics,
  * (1) compared between PD freezers whose FOG responds to SCS and those whose FOG does not respond to SCS (in all 29 patients of the intervention group, at the end of the trial stimulation).
  * (2) Compared between on- and off medication state, and between DBS-on and DBS-off state (in PD freezers from the intervention group who received a permanent SCS implant, at 6 month follow-up; and in control group 2).
  * (3) compared between PD freezers (from the intervention group who received a permanent SCS implant, at 6 month follow-up), SCS patients without PD (control group 1) and SCS patients with PD but without FOG (control group 2).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe De Vloo, MD, PhD, Prof., Principal Investigator — Department of Neurosurgery, University Hospitals Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided